CLINICAL TRIAL: NCT06027645
Title: Effects of Early Crawling Training Via a Mini-Skateboard on the Motor Development of Very Premature Infants at Risk For Neurodevelopmental Disorder
Brief Title: Early Intervention Based on Neonatal Crawling in Very Premature Infants at Risk For Neurodevelopmental Disorder
Acronym: Premalocom2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marianne Barbu-Roth (Other)
Collaborators: Ecole Pratique des Hautes Etudes (Other); Université Paris Cité (Other); San Francisco State University (Other); Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor-Investigator, Marianne Barbu-Roth, Principal Investigator, Centre National de la Recherche Scientifique, France
Organization: Centre National de la Recherche Scientifique, France (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Premalocom2
Record Dates: First submitted 2023-08-31; First posted 2023-09-07 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Prematurity; Extreme Prematurity; Infant Development; Brain Damage; Motor and Developmental Delay
Keywords: Prematurity; Crawling; Early intervention; Motor development; Locomotion
MeSH Terms: conditions — Premature Birth; Brain Injuries; Learning Disabilities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Crawli Group (Experimental): Participants from the Crawli Group will benefit from the crawling stimulation intervention with a mini-skateboard (i.e. the crawliskate) in addition to usual care
  Interventions: Behavioral: Crawling stimulation with a mini-skateboard (i.e. the crawliskate)
- Control Group (No Intervention): Control group infants benefit from usual care

INTERVENTIONS:
Behavioral: Crawling stimulation with a mini-skateboard (i.e. the crawliskate) — Consists of 8 weeks of daily training. Infants benefit from a 10 minutes session everyday at home with either a trained therapist or his/her parents. Parents are trained by the therapist at the begining of the 8 weeks. During each session the infant is prone wrapped on a mini-skateboard (i.e. the crawliskate) and has to produce flexion and extension movements with his four limbs in order to move forward with the assistance of the adult (therapist or parent).
  Arms: Crawli Group

SUMMARY:
Extreme prematurity is constantly increasing according to the World Health Organization. However, methods to train premature infants at risk of disability is sorely lacking. The goal of this project is to overcome this problem. In previous studies, the investigators discovered that promoting the crawling of typical newborns on a mini skateboard, the Crawliskate (a new tool that the investigators designed and patented EP2974624A1), is an excellent way to stimulate infants' motor and locomotor development. This method is a promising way to provide early interventions in infants at heightened risk for developmental delay, such as premature infants.

The specific objective of this study is to determine if early training in crawling on this mini skateboard will accelerate motor (particularly locomotor) and/or neuropsychological development in very premature infants identified as high risk for developmental delay.

Methodology: The investigators will study and follow two groups of very premature infants born between 24 and 26 weeks of gestational age or born between 26 and 32 with major brain lesions.

These infants will be recruited before their hospital discharge at the NICU. After their discharge from the hospital, one group of infants will be trained at home by their parents under the supervision of physiotherapists to crawl on the Crawliskate every day for 2 months (Crawli group), and one group of infants will receive regular medical care (Control group). All infants will be tested for: 1)their crawling proficiency on the Crawliskate at term-equivalent age (just before training for the trained groups) and at 2 and 6 months corrected age (CA, i.e., age determined from the date on which they should have been born), 2) their motor proficiency between 2 and 12 months CA (2D and 3D recording of head control, sitting, crawling, stepping, walking) and 3) their neurodevelopmental, motor and neuropsychological development between 0 and 28 months CA: BSID III edition, ASQ-3, Amiel-Tison's Neurological Assessment, Prechtl Assessment of general movements. One more ASQ-3 questionnaire will be provided at five years.

Expected results: The first research hypothesis is that premature infants trained daily to crawl (for two months after discharge from the NICU) will acquire proficient crawling patterns and develop earlier and more effective motor and neuropsychological development than premature infants who receive no training.

ELIGIBILITY:
Inclusion Criteria:

* Term between 24-26 GA or 26-32 GA with suspected brain lesion
* parental consent
* family living in intervention area
* good tolerance on the first crawliskate trial

Exclusion Criteria:

* no bronchodysplasia defined by oxygen dependency after 36 GA
* no medical disease
* no limb deformity
* no karyotype anomaly
* no visual or auditory impairment

Ages: 39 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2021-03-29 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Gross motor score from the Bayley Scale of Infant and toddlers Development III ed. | 12 months corrected age
  The Bayley Scale of Infant and toddlers Development III ed. (BSID III) assesses several aspect of development: motor, fine motor, communication, personal social, language and problem solving domain.
  A score can be obtained for each aspect. At 12 months corrected age we only evaluate gross and fine motor scores, and we consider the gross motor score obtained at 12 months corrected age as the primary outcome of our study.
  The minimal score is 0 and there is no maximal score (the child is asked to complete several tasks, and the test can continues with questions from an upper age and only stops when a child no longer succeed with the tasks to complete). A higher score means more advanced skills.

SECONDARY OUTCOMES:
Amiel-Tison Neurological Assessment | at 39-42 gestational age, 2, 9, 12 months corrected age
  Infant neurological examination at study entry and after the training
Prechtl assessment | at 39-42 gestational age and 2 months corrected age
  General movements assessment by video recording: measures the fluency and variability of spontaneous movement while the infant is lying supine on a mattress
Age and Stage questionnaire (ASQ) 3 | 2, 6, 9, 12, 18, 28 corrected age and 5 years
  Parental appreciation of their infant development in personal-social, communication, gross motor, fine motor and problem solving domain The minimal score is 0 and the maximal score is 60. A higher score means more advanced skills.
2D & 3D analysis of movement | at 39-42 gestational age, 2, 6, 9, 12 months corrected age
  2D & 3D analysis of movement (head control, sitting, crawling, stepping, walking) using a motion capture system.
Fine and gross motor scores from the Bayley Scale of Infant and toddlers development III ed. | 2, 6, 9, 12, 24 months corrected age
  The Bayley Scale of Infant and toddlers Development III ed. (BSID III) assesses several aspect of development: motor, fine motor, communication, personal social, language and problem solving domain.
  A score can be obtained for each aspect. At 2, 6, 9, 12 and 24 months corrected age we only evaluate fine and gross motor scores. Note that the gross motor score obtained at 12 months corrected age is the primary outcome of our study but the fine motor score obtained at 12 months corrected age is also a secondary outcome.
  The minimal score is 0 and there is no maximal score (the child is asked to complete several tasks, and the test can continues with questions from an upper age and only stops when a child no longer succeed with the tasks to complete). A higher score means more advanced skills.

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Barbu-Roth, PhD, Study Chair — Centre National de la Recherche Scientifique, France; Valérie Biran, MD, PhD, Principal Investigator — APHP
Locations (3):
- France (3):
  - Hôpital Paris Saint-Joseph, Paris
  - Cnrs Umr 8002, Paris, Île-de-France Region
  - Hôpital Robert Debré, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: Yes
IPD will be made available upon reasonable request to corresponding author
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: From 2025 to 2030
Access Criteria: IPD will be made available upon reasonable request to corresponding author